CLINICAL TRIAL: NCT02912299
Title: Onderzoek Naar Intracutane Natriumopslag Bij Intensive Care patiënten (InCa-studie)
Brief Title: Investigation on Differences in Skin Sodium Content Between Normal Subjects and ICU-patients
Acronym: InCa
Status: Completed | Type: Observational
Sponsor: Frisius Medisch Centrum (Other)
Collaborators: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: NL 56729.099.16
Record Dates: First submitted 2016-09-13; First posted 2016-09-23 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Hypernatremia
MeSH Terms: conditions — Hypernatremia | interventions — Blood Specimen Collection; Urinalysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Slides for microscopic investigations, containing slices of the skin biopsies. These biopsies are only diagnostic and these are specific and only for study properties. Study involvement will not influence diagnostic or therapeutic interventions that are due to common treatment.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Septic patients: Patients admitted to the ICU that fulfill the criteria for the systemic inflammatory response syndrome in the presence of a(n expected) new infection. 2 3mm skin biopsies will be taken, blood and urine analysis will take place and also blood collection for RNA-investigation.
  Interventions: Procedure: Skin biopsies; Other: Blood and urine analysis; Other: Blood collection for RNA-investigation
- CABG patients: Patients admitted to the ICU after coronary artery bypass grafting. 2 3mm skin biopsies will be taken, blood and urine analysis will take place and also blood collection for RNA-investigation.
  Interventions: Procedure: Skin biopsies; Other: Blood and urine analysis; Other: Blood collection for RNA-investigation
- Patients before hip replacement: Patients that will undergo a hip replacement because of arthrosis. 2 3mm skin biopsies will be taken, blood and urine analysis will take place and also blood collection for RNA-investigation.
  Interventions: Procedure: Skin biopsies; Other: Blood and urine analysis; Other: Blood collection for RNA-investigation

INTERVENTIONS:
Procedure: Skin biopsies — 2 3mm skin biopsies will be taken
Other: Blood and urine analysis — Measurement of sodium, potassium and kidneyfunction in blood and urine.
Other: Blood collection for RNA-investigation — A blood sample that, in case of relevant differences between groups, could be used for RNA-profiling.

SUMMARY:
This study investigates the differens in sodium storage in skin between normal subjects, patients after cardiac surgery and septic patients.

DETAILED DESCRIPTION:
According to the current paradigm ICU-acquired hypernatremia is mainly an iatrogenic problem, caused by sodium overload or water deficit. In spite of several interventions to reduce sodium intake and optimize fluid balance, critically ill patients still develop hypernatremia. These patients also seem to have an inability to excrete sodium, hence develop a positive sodium balance. In animals sodium storage in the third compartment was found. Our hypothesis is that sodium storage in the third compartment is different in critically ill patients and this difference could play a role in the development of ICU-acquired hypernatremia.

ELIGIBILITY:
Inclusion Criteria:

* 50-80 years (septic patients), 45-85 years (CABG and hip replacement-patients)
* Patients undergoing hip replacement: no relevant medical history (i.e. chronic and/or systemic diseases with a suspected influence on sodium / sodium handling)
* Septic patients: fulfilling the criteria for the systemic inflammatory response syndrome in the presence of a(n expected) new infection

Exclusion Criteria:

* Absence of both upper legs
* Skin disease that makes skin biopsies in healthy skin impossible
* Subjects with in their history formation of exaggerated scar tissue
* Subjects suffering from psoriasis or lichen ruber
* Use of skin corticosteroids on all skin of both upper legs < 2 weeks before inclusion
* Tattoos covering the whole surface of both upper legs
* Use of diuretics in the past month
* Current renal replacement therapy
* Septic patients: not being sedated
* Patients undergoing hip replacement: hip replacement because of an inflammatory disease

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * 15 patients admitted to the ICU with systemic inflammatory response syndrom in the presence of a(n expected) new infection
  * 15 patients admitted to the ICU after coronary artery bypass surgery, matched by gender and age (+/- 10 years) to the septic patients
  * 15 patients undergoing a hip replacement for arthrosis, matched by gender and age (+/- 10 years) to the septic patients
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2017-09-05 (Actual); Study Completion 2017-09-05 (Actual)

PRIMARY OUTCOMES:
Difference in sodium concentration in skin biopsy between groups | Different for the separate groups: before hip replacement, within 2 hours after CABG and within 12 hours after admission for septic patients
  Skin biopsies will be taken within the described time frame, analysis will take place after all biopsies of all subjects are included

SECONDARY OUTCOMES:
Immunohistochemistry: outcomes of proteoglycans | Different for the separate groups: before hip replacement, within 2 hours after CABG and within 12 hours after admission for septic patients
Immunohistochemistry: binding capacity of proteoglycans | Different for the separate groups: before hip replacement, within 2 hours after CABG and within 12 hours after admission for septic patients
Immunohistochemistry: density of lymph capillaries | Different for the separate groups: before hip replacement, within 2 hours after CABG and within 12 hours after admission for septic patients
Immunohistochemistry: presence of macrophage influx | Different for the separate groups: before hip replacement, within 2 hours after CABG and within 12 hours after admission for septic patients
Quantification of different matrix components / proteoglycans: decorine - if enough tissue is available | Different for the separate groups: before hip replacement, within 2 hours after CABG and within 12 hours after admission for septic patients
Quantification of different matrix components / proteoglycans: versican (if enough tissue is available) | Different for the separate groups: before hip replacement, within 2 hours after CABG and within 12 hours after admission for septic patients
Quantification of different matrix components / proteoglycans: biglycan- if enough tissue is available | Different for the separate groups: before hip replacement, within 2 hours after CABG and within 12 hours after admission for septic patients
mRNA profiling of proteoglycans and synthesizing enzymes by way of RNA-isolation - if enough tissue is available | Different for the separate groups: before hip replacement, within 2 hours after CABG and within 12 hours after admission for septic patients

CONTACTS AND LOCATIONS:
Overall Officials: Christiaan Boerma, MD PhD, Principal Investigator — medical center leeuwarden; Jaap van den Born, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- Medisch Centrum Leeuwarden, Leeuwarden, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Depending on the requests of the magazine involved.

REFERENCES:
- [Background] Polderman KH, Schreuder WO, Strack van Schijndel RJ, Thijs LG. Hypernatremia in the intensive care unit: an indicator of quality of care? Crit Care Med. 1999 Jun;27(6):1105-8. doi: 10.1097/00003246-199906000-00029. PMID 10397213
- [Background] Waite MD, Fuhrman SA, Badawi O, Zuckerman IH, Franey CS. Intensive care unit-acquired hypernatremia is an independent predictor of increased mortality and length of stay. J Crit Care. 2013 Aug;28(4):405-12. doi: 10.1016/j.jcrc.2012.11.013. Epub 2013 Jan 29. PMID 23369520
- [Background] Lee JW. Fluid and electrolyte disturbances in critically ill patients. Electrolyte Blood Press. 2010 Dec;8(2):72-81. doi: 10.5049/EBP.2010.8.2.72. Epub 2010 Dec 31. PMID 21468200
- [Background] Titze J, Krause H, Hecht H, Dietsch P, Rittweger J, Lang R, Kirsch KA, Hilgers KF. Reduced osmotically inactive Na storage capacity and hypertension in the Dahl model. Am J Physiol Renal Physiol. 2002 Jul;283(1):F134-41. doi: 10.1152/ajprenal.00323.2001. PMID 12060595
- [Background] Titze J, Lang R, Ilies C, Schwind KH, Kirsch KA, Dietsch P, Luft FC, Hilgers KF. Osmotically inactive skin Na+ storage in rats. Am J Physiol Renal Physiol. 2003 Dec;285(6):F1108-17. doi: 10.1152/ajprenal.00200.2003. Epub 2003 Jul 29. PMID 12888617